CLINICAL TRIAL: NCT05679050
Title: Single-arm, Single-centered, Open-label Phase II Study on Sequential AG Regimen and FOLFIRINOX Regimen as Neoadjuvant Therapy in Patients With Resectable Pancreatic Cancer
Brief Title: Phase II Study on Sequential AG and FOLFIRINOX as Neoadjuvant Therapy in Patients With Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJGI-005
Record Dates: First submitted 2022-11-15; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-11

CONDITIONS: Resectable Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AG Regimen Followed by FOLFIRINOX Regimen (Experimental): AG Regimen Followed by FOLFIRINOX Regimen
  Interventions: Drug: AG Followed by FOLFIRINOX

INTERVENTIONS:
Drug: AG Followed by FOLFIRINOX — AG（every 28 days) Nab-paclitaxel 125 mg/m2 i.v. over 30 min, gemcitabine hydrochloride 1g/m2 i.v. over 30 min, D1, 8 and 15 ; FOLFIRINOX(every 42 days) Oxaliplatin: 65 mg/m2 i.v. over 2h on D1, 15, 29; Tetrahydrofolate: 400 mg/m2 i.v.2h on D1, 15, 29; Irinotecan: 150 mg/m2 i.v. over 90 min every 42 days on D1, 15, 29; 5-FU: 2400 mg/m2 i.v. over 46h /14 days on D1-3, 15-17, and 29-31; After one round of above therapy, patients achieving stable disease and above without disease progression or unacceptable toxicity underwent pancreatectomy within 4-8 weeks; Patients who did not achieve stable disease and above were treated another round , and patients who achieved stable disease and above underwent pancreatectomy at 4-8 weeks.
  Following pancreatectomy, patients underwent AG regimen (2 rounds, 56 days) followed by FOLFIRINOX regimen (42 days) in the absence of disease progression or unacceptable toxicity, and AG and FOLFIRINOX dosing as the preoperative therapy.

SUMMARY:
Based on the safety and benefit of neoadjuvant therapy for patients with pancreatic cancer in the available evidence, as well as the principle of sequential chemotherapy with different regimens and the existing preliminary investigation , the aim of this study was to further explore the efficacy and safety of neoadjuvant therapy with AG regimen followed by FOLFIRINOX regimen in patients with resectable pancreatic cancer, and to assess the impact of neoadjuvant therapy on the health-related quality of life of patients, in order to bring new treatment options for neoadjuvant therapy of pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is known as the king of cancer and is one of the malignant tumors with a very high mortality rate in the digestive system, which is characterized by a high degree of malignancy and a poor prognosis. The current standard of care is surgical resection followed by adjuvant therapy. However, patients treated with standard surgery had a 2-year median overall survival of approximately 40%. Neoadjuvant therapy can reduce the tumor to a certain extent and downstage the tumor, so as to achieve more R0 resection, reduce the postoperative recurrence rate and prolong survival.

SWOG S1505 published by ASCO in 2020 demonstrated adequate safety and high resectability rates for perioperative chemotherapy. The study concluded that perioperative chemotherapy has adequate safety and a high resectability rate. However, neither regimen in this study demonstrated an improvement in OS compared with prior standard therapies. Neoadjuvant treatment of pancreatic cancer therefore remains a long way to go.

Recent results from the NEONAX perioperative randomized phase II study for pancreatic cancer presented at the ASCO meeting in 2022 confirmed the benefit of neoadjuvant therapy and demonstrated the OS benefit brought about by neoadjuvant therapy.

Neoadjuvant regimens require regimens with good tumor shrinkage and high response rate, and there is no standard regimen for neoadjuvant therapy of pancreatic cancer, often referring to regimens with high response rate for advanced treatment. However, due to the high malignancy and disease particularity of pancreatic cancer, there is no advanced treatment regimen with high response rate. The mFOLFIRINOX (5-fluorouracil, irinotecan, oxaliplatin) and AG regimens (gemcitabine combined with nab-paclitaxel) are commonly used regimens in clinical practice. Therapeutic options for pancreatic cancer are limited, therefore, different combinations and application sequences of existing regimens are one of the directions explored in clinical research.

In summary, based on the safety and benefit of neoadjuvant therapy for patients with pancreatic cancer in the available evidence, as well as the principle of sequential chemotherapy with different regimens and the existing preliminary study exploration, the aim of this study was to further explore the efficacy and safety of neoadjuvant therapy with AG regimen followed by FOLFIRINOX regimen in patients with resectable pancreatic cancer, and to assess the impact of neoadjuvant therapy on the health-related quality of life of patients, in order to bring new treatment options for neoadjuvant therapy of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed pancreatic cancer.
2. ECOG performance status must be 0-1.
3. 18-75 years
4. patients must have measurable pancreatic disease. CT scans or MRIs to assess measurable disease must have been completed within 28 days prior to enrollment. All disease must be assessed and documented on the Baseline Tumor Assessment form.
5. Patients must have a primary tumor resectable on contrast-enhanced CT or MRI of the chest, abdomen, and pelvis, which is defined as: (1) no involvement of the celiac artery, common hepatic artery, and superior mesenteric artery. (2) The portal vein and/or superior mesenteric vein were not involved, or the interface between the tumor and the vessel wall was < 180 °; the portal vein/splenic vein confluence was patent. (3) No evidence of metastatic disease. Lymphadenopathy outside the operative pelvis (defined as lymph nodes with a short axis > 1 cm) (ie, para-aortic, pericaval, celiac trunk, or distal lymph nodes) was considered M1 disease, rendering the patient ineligible. However, if these lymph nodes are biopsied and negative, enrollment may be considered following review by the study chair. Note: For pancreatic body and tail tumors, any degree of splenic arteriovenous involvement is considered resectable.
6. Patients must receive surgical consultation within 21 days before registration to verify whether the patient is eligible for surgery;
7. Patients must have normal hematological function within 14 days before registration, including: ANC > 1,500/mcL; platelets > 100,000/mcL; hemoglobin > 9 g/dL.
8. Patients must have normal liver function within 14 days prior to enrollment as evidenced by: total bilirubin < 1.5 × upper limit of normal (1ULN); AST and ALT < 3 × 1ULN; serum albumin > 3 g/dL.
9. Patients must have normal renal function as indicated by serum creatinine ≤ 1 ULN within 14 days prior to enrollment.

Exclusion Criteria:

1. Previous surgery, radiotherapy, chemotherapy, targeted therapy, or any investigational therapy for pancreatic cancer.
2. Histology other than adenocarcinoma or any mixed histological features.
3. Patients with uncontrolled concurrent medical conditions including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements were excluded.
4. No prior malignancy is allowed except for adequately treated basal (or squamous) skin cancer, in situ cervical cancer, in situ breast cancer (ductal or lobular). Tumors were eligible if they were eradicated and had no evidence of disease for more than 3 years.
5. Patients must not be pregnant or breastfeeding because there is a risk of harm to the fetus or nursing infant. Females/males of childbearing potential must agree to use an effective method of contraception for 3 months following the last dose of chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | Within 4-8 weeks of last dose of pre-operative chemotherapy
  Percentage of patients who achieved R0 resection
Disease-free Survival(DFS) | 4 years
  Duration of patients alive without recurrence of disease

SECONDARY OUTCOMES:
Operation Rate | Within 4-8 weeks of last dose of pre-operative chemotherapy
  Percentage of patients who complete operation
Objective Response Rate | Within 4-8 weeks of last dose of pre-operative chemotherapy
  Percentage of patients who achieved partial response or complete response
2-year Overall Survival Rate | from treatment initiation until death due to any cause, assessed up to 2 year
  Percentage of patients alive at two years
Local or distant recurrence after R0 or R1 resection Rates | 4 years
  Percentage of patients who have Local or distant recurrence after R0 or R1 resection Rates
Treatment-Emergent Adverse Event Rate | 1 year
  Percentage of TEAE

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Liu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No